CLINICAL TRIAL: NCT00602511
Title: Thalidomide Versus Bortezomib in Melphalan Refractory Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Myeloma Study Group (Other)
Responsible Party: Martin Hjorth, Department of Medicine, Lidköping Hospital, S-53185 Lidköping, Sweden
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NMSG 17/07; EudraCT no. 2007-001292-11
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Multiple Myeloma
Keywords: Melfalan refractory multiple myeloma; Multiple myeloma; Relapsing; Refractory; Thalidomide; Bortezomib; Randomized clinical trial
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Bortezomib - dexamethasone
  Interventions: Drug: Bortezomib
- 2 (Experimental): Thalidomide - dexamethasone
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1,3 mg/m2 intravenously on days 1, 4, 8 och 11 of every 3 weeks cycle until maximal response, toxicity or maximum 8 cycles
  Dexamethasone 20 mg days 1-2, 4-5, 8-9 and 11-12 during the first 2 cycles, thereafter individualized dose depending on response and toxicity
  Arms: 1
Drug: Thalidomide — Thalidomide 50 mg/day with dose escalation every 3 weeks until response or toxicity, maximal dose 200 mg/day
  Dexamethasone 40 mg/day day 1-4 every 3 weeks for at least 2 courses, thereafter individualized dose depending on response and toxicity
  Arms: 2

SUMMARY:
The purpose of the study is to compare thalidomide + dexamethasone with bortezomib + dexamethasone in patients with multiple myeloma refractory to melphalan therapy. The main goal is to find out which of these two 2:nd line regimens that offers the patients the best chance for a response with as long duration and as good quality of life as possible.

DETAILED DESCRIPTION:
The study is an open randomized multicentre study in which patients with multiple myeloma refractory to melphalan therapy are randomized between bortezomib and thalidomide therapy, in both arms with the addition of dexamethasone. In case of failure to the initially given treatment the patient will be crossed over to the alternative treatment.

The number of patients needed is calculated to 300, based upon the hypothesis of a 50% difference in progression free survival, a significance level of 95% and a power of 80%. With 12 patients being recruited each month during 25 months and a 4 months follow-up after the last included patient, the total study time will be 29 months.

The dose regimens for bortezomib and thalidomide follow general clinical praxis as regards recommendations for optimal dosing in the Nordic countries.

Evaluation of response and toxicity is performed every 3 weeks for at least 12 weeks, thereafter every 6 weeks. Evaluation of efficacy is done according to The International Myeloma Working Group Uniform Response Criteria. Evaluation of toxicity is done by CTCAE grading. Evaluation of quality of life is done by the EORTC QLQ30 questionnaires with the addition of the myeloma specific MY-24 module which are mailed to the patients at predetermined intervals during the study.

ELIGIBILITY:
Inclusion Criteria:

* Treatment demanding multiple myeloma
* Refractoriness to melphalan
* Acceptance of rules for prevention of pregnancy

Exclusion Criteria:

* Previous treatment with bortezomib, thalidomide, or lenalidomide
* Sensory neuropathy grade III or neuropathic pain grade II
* Severe concomitant disorder, e.g. other malignancy or severe heart disease
* Transformation to plasma cell leukemia or aggressive lymphoma
* Frequent visits for bortezomib injections not feasible
* Anticipated non-adherence to study protocol
* Pregnancy
* Anticipated non-adherence to rules for prevention of pregnancy
* Severe thrombocytopenia (Thrombocyte count less than 25000/microliter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival

SECONDARY OUTCOMES:
Response rate
Response duration
Time to start of other treatment
Toxicity
Quality of life
Response rate after cross-over
Response duration after cross-over

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hjorth, MD, PhD, Principal Investigator — Department of Medicine, Lidköping Hospital, S-53185 Lidköping, Sweden
Locations (27):
- Denmark (5):
  - Ålborg university Hospital, Aalborg
  - Århus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev University Hospital, Herlev
  - Odense University Hospital, Odense
- Norway (4):
  - Ullevål Sykehus, Oslo
  - Diakonhjemmet, Oslo
  - Stavanger Universitetssykehus, Stavanger
  - Trondheim University Hospital, Trondheim
- Sweden (18):
  - Falun Hospital, Falun
  - Gävle Hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborg Hospital, Helsingborg
  - Lidköping Hospital, Lidköping
  - Lund University Hospital, Lund
  - Malmö University Hospital, Malmo
  - Mölndal hospital, Mölndal
  - Örebro University Hospital, Örebro
  - Örnsköldsvik Hospital, Örnsköldsvik
  - Skövde Hospital, Skövde
  - St Göran Hospital, Stockholm
  - Sundsvall Hospital, Sundsvall
  - Uddevalla Hospital, Uddevalla
  - Norrland University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
  - Växjö Hospital, Vaxjo
  - Västerås Hospital, Västerås